CLINICAL TRIAL: NCT04703699
Title: A Retrospective, Multinational, Multicentre, Observational Study in Patients Presenting With Native Severe Aortic Valve Stenosis and Treated With Myval™ Transcatheter Heart Valve Series in Real-world Setting.
Brief Title: Myval Global Study of Myval™ THV Series Implanted in Patients With Native Severe Aortic Valve Stenosis.
Status: Recruiting | Type: Observational
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MLS/MYV-3/Global study
Record Dates: First submitted 2020-12-22; First posted 2021-01-11 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Myval Transcatheter Heart Valve Series — Myval™ THV is a newer-generation balloon-expandable THV characterized by a nickel-cobalt alloy frame composed of a single element - hexagon arranged in a hybrid honeycomb fashion.
  Other Names: Myval THV

SUMMARY:
A retrospective, multinational, multicentre, observational study in patients presenting with native severe aortic valve stenosis and treated with Myval™ Transcatheter Heart Valve Series in real-world setting.

DETAILED DESCRIPTION:
Myval Global Study: A retrospective, multicentre, observational study in patients presenting with native severe aortic valve stenosis and treated with Myval™ Transcatheter Heart Valve Series in real-world setting.

This study shall retrospectively collect the data of minimal 200 consecutive patients treated with Myval™ THV Series approximately 15 participating sites Globally.

Primary Endpoint:

Primary Combined Safety and Effectiveness Endpoint: [Time frame: 30 days]

It is the composite of following:

* All-cause mortality
* All stroke
* Bleeding (type 3 and 4)
* Acute kidney injury (stage 2 ,3 & 4)
* Major vascular complications
* Moderate or severe prosthetic valve regurgitation
* Conduction system disturbances resulting in a new permanent pacemaker implantation.

Secondary endpoints:

1. All-cause mortality (VARC-3 defined criteria) [Time Frame: Through 30 days]
2. All stroke (VARC-3 defined criteria) [Time Frame: Through 30 days]
3. Acute Kidney Injury (AKI) based on the Acute Kidney Injury Network (AKIN) System Stage 2, Stage 3 or Stage 4 [Time Frame: Through 30 days]
4. Bleeding type 3 and 4 (VARC-3 criteria) [Time Frame: Through 30 days]
5. Moderate or severe prosthetic valve regurgitation [Time Frame: Through 30 days]
6. New permanent pacemaker implantation [Time Frame: Through 30 days] New permanent pacemaker implantation rates will be analyzed further based on the patient's history of left and/or right bundle branch block.
7. Conduction disturbances and arrhythmias according to VARC-3 [Time Frame: Through 30 days]
8. Device success (VARC-3 criteria) [Time Frame: Pre-discharge]
9. Early safety at 30 days (VARC-3 criteria) [Time Frame: After 30 days of index procedure]
10. Clinical efficacy after 30 days (VARC-2 criteria) [Time Frame: After 30 days of index procedure]
11. Time-related valve safety (VARC-2 criteria) [Time Frame: Through 30 days]
12. Vascular and access related complications (VARC-3 criteria) [Time Frame: Pre-discharge, Through 30 days]
13. Major vascular complications (VARC-3 criteria) [Time Frame: Pre-discharge, Through 30 days]
14. Functional improvement from baseline as measured per

    a. NYHA functional classification [Time frame: Baseline, 30 days]
15. Echocardiographic End Points

    * Effective orifice area (EOA)
    * Index effective orifice area (iEOA)
    * Mean aortic valve gradient
    * Peak aortic valve gradient
    * Peak aortic velocity
    * Transvalvular, paravalvular and total aortic regurgitation
    * Left ventricular ejection fraction (LVEF)
    * Valve calcification
    * Cardiac output and cardiac index [Time frame: Through 30 days]
16. Patient-prosthesis Mismatch: [Time Frame: Post-procedure, predishcarge, Through 30 days] Severity patient-prosthesis-mismatch will be based on following

    * For subjects with BMI < 30 kg/m2, index effective orifice area (EOAi) 0.85 - 0.66 cm2 /m2 for moderate and ≤0.65 cm2 /m2 for severe
    * For subjects with BMI ≥30 kg/m2, index effective orifice area (EOAi) 0.70 - 0.56 cm2 /m2 for moderate and ≤0.55 cm2 /m2 for severe BMI = weight(kg)/(height (m)) 2
17. Length of index hospital stay. [Time frame: At discharge]

    - Number of days from hospital admission to discharge.
18. Re-hospitalization (VARC-3 defined criteria) [Time Frame: Through 30 days]
19. New onset of atrial fibrillation or atrial flutter [Time Frame: Post-procedure, Pre-discharge and 30 days]
20. Endocarditis [Time Frame: Through 30 days]
21. Major bleeding event [Time Frame: Through 30 days]
22. Other Endpoints:

    * Myocardial rupture [Time Frame: During procedure]
    * Paravalvular leak [Time Frame:Through 30 days]
    * Degree of over- or under-expansion of Myval [Time Frame: During procedure]
    * Accuracy of deployment in relation to the annular plane [Time Frame: During procedure]
    * Pacemaker deployment (and the symptoms resulting in it) [Time Frame: Through 30 days]
    * Interference with the mitral valve; and [Time Frame: During procedure]
    * Interference with the LVOT [Time Frame: During procedure]

      * If the endpoint data is available through 1 year, it will also be collected and analyzed.

Clinical efficacy data will be collected only for patients with availability of data after 30 days follow-up.

Long term clinical follow up by telephonic interview will be conducted for all patients who have completed 30 days safety follow-up, at 1 year, 3 year and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients of this study must have received Myval™ THV series for treatment of native severe aortic stenosis and completed a minimum of 30-day follow-up.

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have been treated with Myval™ THV series will be selected for the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Effectiveness as defined by the Valve Academic Research Consortium-3 (VARC-3) | 30 day
  It is the composite of following
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening or disabling bleeding
  * Acute kidney injury (stage 2 or 3)
  * Major vascular complications
  * Moderate or severe prosthetic valve regurgitation
  * Conduction system disturbances resulting in a new permanent pacemaker implantation

SECONDARY OUTCOMES:
All-cause mortality | 30 day
  Number of mortality as per VARC - 3 Criteria
All stroke | Through 30 days
Acute Kidney Injury (AKI) based on the Acute Kidney Injury Network (AKIN) System Stage 2, Stage 3 or Stage 4 | Through 30 days
  Number of participants of AKI as per AKIN Network
Bleeding type 3 and 4 | Through 30 days
  Number of participants for bleeding as per VARC-3 criteria
Moderate or severe prosthetic valve regurgitation | Through 30 days
New permanent pacemaker implantation | Through 30 days
  New permanent pacemaker implantation rates will be analyzed further based on the patient's history of left and/or right bundle branch block
Conduction disturbances and arrhythmias | Through 30 days
  Number of participants for Conduction disturbances and arrhythmias as per VARC-3 Criteria
Device Success | During hospital stay or maximum of 7 days after index procedure, whichever is earlier.
  Number of participants for Device success as per VARC-3 Criteria
Early safety at 30 days | After 30 days of index procedure
  Number of participants for Early safety as per VARC-3 Criteria
Clinical efficacy after 30 days | After 30 days of index procedure
  Number of participants for Clinical efficacy as per VARC-2 Criteria
Time related valve safety | Through 30 days
  Number of participants for Time related valve safety as per VARC-2 Criteria
Vascular and access related complications | Pre-discharge, Through 30 days
  Number of participants for Vascular and access related complications as per VARC-3 Criteria
Major vascular complications | Pre-discharge, Through 30 days
  Number of participants for Major vascular complications as per VARC-3 Criteria
Functional improvement from baseline as measured | Baseline, 30 days
  Number of participants for Functional improvement as per NYHA functional classification
Echocardiographic End Points | Through 30 days]
  * Effective orifice area (EOA)
  * Index effective orifice area (iEOA)
  * Mean aortic valve gradient
  * Peak aortic valve gradient
  * Peak aortic velocity
  * Transvalvular, paravalvular and total aortic regurgitation
  * Left ventricular ejection fraction (LVEF)
  * Valve calcification
  * Cardiac output and cardiac index
Patient-prosthesis Mismatch | Through 30 days
  Severity patient-prosthesis-mismatch will be based on following For subjects with BMI < 30 kg/m2, index effective orifice area (EOAi) 0.85 - 0.66 cm2/m2 for moderate and ≤0.65 cm2/m2 for severe For subjects with BMI ≥30 kg/m2, index effective orifice area (EOAi) 0.70 - 0.56 cm2 /m2 for moderate and ≤0.55 cm2/m2 for severe BMI = weight(kg)/(height (m)) 2
Length of index hospital stay | At discharge
  Number of days from hospital admission to discharge
Re-hospitalization | Through 30 days
  Number of participants as per VARC-3 defined criteria
New onset of atrial fibrillation or atrial flutter | Post-procedure, Pre-discharge and 30 days
  VARC-3 criteria
Endocarditis | Through 30 days
  Number of participants for Endocarditis as per VARC-3 criteria
Major bleeding event | Through 30 days
  Number of participants for Major bleeding event as per VARC-3 criteria
Myocardial rupture | During procedure
  Number of participants for Myocardial rupture
Paravalvular Leak | Through 30 days
  Number of participants for Paravalvular Leak
Degree of over - or Under-expansion of Myval | During Procedure
  Number of participants for Degree of over - or Under-expansion of Myval
Accuracy of deployment in relation to the annular plane | During procedure
  Number of participants for Accuracy of deployment in relation to the annular plane
Pacemaker deployment (and the symptoms resulting in it) | Through 30 days
  Number of participants for Pacemaker deployment (and the symptoms resulting in it)
Interference with the mitral valve | During procedure
  Number of participants for Interference with the mitral valve
Interference with the LVOT | During procedure
  Number of participants for Interference with the LVOT

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Thakkar, Ph.D., Study Chair — Head - Clinical Research and Medical Writing
Locations (8):
- North Estonia Medical center, Tallinn, Estonia
- Clinical Institute Saint Ambrogio, Milan, Italy
- Amphia Ziekenhui, Breda, North Brabant, Netherlands
- University of Gdansk, Gdansk, Bażyńskiego, Poland
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Spain (2):
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Cliinico Univertistario de Valladolid, Valladolid
- Kocaeli University School of Medicine, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No